CLINICAL TRIAL: NCT06572280
Title: Non-invasive Phrenic Nerve Stimulation in ARDS Patients - a Feasibility Study
Brief Title: Non-invasive Phrenic Nerve Stimulation in ARDS Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NPES-diaphragm protection
Record Dates: First submitted 2024-08-14; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: ARDS, Human; Ventilator-Induced Lung Injury; Diaphragm Injury
Keywords: ARDS; diaphragm injury; mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNS group (Experimental): Electrical stimulation of the phrenic nerve in ARDS patients.
  Interventions: Device: PNS group

INTERVENTIONS:
Device: PNS group — non-invasive phrenic nerve stimulation

SUMMARY:
Reduced diaphragmatic activity during mechanical ventilation can lead to diaphragmatic disuse atrophy, atelectasis, increased lung stress and strain, and hemodynamic impairment. This, in turn, may prolong the duration of mechanical ventilation, make weaning more difficult, and even increase mortality. Synchronizing phrenic nerve stimulation to promote diaphragmatic activity may prevent ventilator-induced lung injury and ventilator-induced diaphragm dysfunction, thereby improving patient outcomes. Surgically implanted phrenic nerve stimulation has been used in certain neurological disorders, but the effects of percutaneous non-invasive synchronized phrenic nerve stimulation in patients with ARDS undergoing mechanical ventilation remain unclear and require further investigation.

DETAILED DESCRIPTION:
Mechanical ventilation is an important treatment for patients with acute hypoxemic respiratory failure (AHRF). However, reduced diaphragmatic activity during mechanical ventilation can lead to diaphragmatic disuse atrophy, atelectasis, increased lung stress and strain, and hemodynamic impairment. This, in turn, may prolong the duration of mechanical ventilation, make weaning more difficult, and even increase mortality in these patients. In patients with AHRF undergoing mechanical ventilation, maintaining moderate spontaneous breathing under lung and diaphragm protective ventilation remains challenging. Synchronizing phrenic nerve stimulation to promote diaphragmatic activity may prevent ventilator-induced lung injury (VILI) and ventilator-induced diaphragm dysfunction (VIDD), thereby improving patient outcomes. Surgically implanted phrenic nerve stimulation has been used in certain neurological disorders, but the effects of percutaneous non-invasive synchronized phrenic nerve stimulation in patients with acute respiratory distress syndrome (ARDS) undergoing mechanical ventilation remain unclear and require further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ARDS patients undergoing controlled mechanical ventilation
2. The duration of endotracheal intubation < 48 hrs

Exclusion Criteria:

1. Neurological condition affecting motor neuron or muscle (e.g. ALS)
2. Paralysis of the phrenic nerve
3. Proven or suspected spinal cord injury
4. Conditions that limit diaphragm movement
5. Patients with Implanted cardiac support systems (pacemaker, implanted defibrillator)
6. Patients with implanted medical pumps
7. Pregnancy
8. Patients with skin lesions, infections or strictures in throat/neck area
9. Patients with metallic implants
10. Refusal to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of enough Tidal volume | Procedure (from enrollment to extubation)
  Percentage of stimulated breaths above the cut-off target tidal volume (3-6 ml/kg ideal body weigh) out of the total number of stimulated breaths
The speed of successful non-invasive electrical stimulation deployment | Procedure (from enrollment to extubation)
  Time between first successful electrical phrenic stimulation and identification of the optimal stimulation locus in seconds

SECONDARY OUTCOMES:
Driving pressure | Procedure (from enrollment to extubation)
  driving pressure was measured in the volume-controlled mode and calculated as the difference between plateau pressure and positive end-expiratory pressure
Diaphragm thickening fraction | up to 28 days
  Diaphragm thickening fraction measured with ultrasound of the diaphragm.
Diaphragm excursion | up to 28 days
  Diaphragm excursion measured with ultrasound of the diaphragm.
Maximal inspiratory pressure (MIP) | Procedure (from enrollment to extubation)
  MIP is measured by the mechanical ventilator during electromagnetic phrenic nerve stimulation.
ventilation distribution | Procedure (from enrollment to extubation)
  ventilation distribution was measured by EIT
Respiratory system compliance | Procedure (from enrollment to extubation)
  Respiratory system compliance is calculated as the ratio of tidal volume to the difference between plateau pressure and positive end-expiratory pressure.

CONTACTS AND LOCATIONS:
Overall Officials: ling liu, phD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No